CLINICAL TRIAL: NCT05752552
Title: A Phase 1 Study to Determine the Safety, and Pharmacokinetics of the Selective MET Kinase Inhibitor, DO-2 in Patients With Advanced or Refractory Solid Tumours
Brief Title: Study to Determine the Safety and Pharmacokinetics of DO-2 in Patients With Advanced or Refractory Solid Tumours
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: DeuterOncology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DO2.22.01
Record Dates: First submitted 2023-02-07; First posted 2023-03-02 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Adult Solid Tumor; Advanced Solid Tumor; Refractory Tumor; Non-small Cell Lung Cancer; Non-small Cell Carcinoma; Lung Cancer; Hereditary Renal Papillary Cancer
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Cohort 1 (starting dose) (Experimental): Oral administration, once a day for 28 days, in a 4-week cycle
  Interventions: Drug: DO-2
- Cohort 2 (dose level 2) (Experimental): Oral administration, once a day for 28 days, in a 4-week cycle
  Interventions: Drug: DO-2
- Cohort 3 (dose level 3) (Experimental): Oral administration, once a day for 28 days, in a 4-week cycle
  Interventions: Drug: DO-2
- Cohort 4 (dose level 4) (Experimental): Oral administration, once a day for 28 days, in a 4-week cycle
  Interventions: Drug: DO-2
- Cohort 5 (dose level 5) (Experimental): Oral administration, once a day for 28 days, in a 4-week cycle
  Interventions: Drug: DO-2
- Cohort 6 (dose level 6) (Experimental): Oral administration, once a day for 28 days, in a 4-week cycle
  Interventions: Drug: DO-2
- Cohort 7 (dose level 7) (Experimental): Oral administration, once a day for 28 days, in a 4-week cycle
  Interventions: Drug: DO-2

INTERVENTIONS:
Drug: DO-2 — Deuterated MET kinase inhibitor

SUMMARY:
This study is a first-in-human, open-label, 2-part, Phase 1 dose escalation study of DO-2, administered orally to patients with advanced or refractory solid tumours, with MET aberrations, and no available, approved therapeutic alternative.

DETAILED DESCRIPTION:
In Part 1, a Simon Design 3 accelerated titration design will be followed. One patient will be enrolled per cohort, until grade 2 toxicity is observed. Three sequential patients per cohort will be enrolled thereafter, with a minimum of 1 week between first dose administration in the first patient and the subsequent ones, in those latter cohorts.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* histologically or cytologically confirmed advanced or refractory solid tumour and no longer eligible for approved, available standard therapies. Tumour types must have:

  1. proven MET activating mutations, determined by previous next generation sequencing (NGS), whole exome sequencing (WES), whole transcriptome sequencing (WTS) or other genomic analysis methods, or
  2. proven amplification (≥ 10 copies) on archived tumour tissue. or
  3. Hereditary Renal Papillary Cancer
* measurable disease in accordance with RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* adequate bone marrow function, without the support of cytokines
* adequate liver function
* adequate renal function
* agree to follow the contraception requirements of the trial
* signed informed consent, indicating study patients understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* major surgery within 3 weeks before enrollment
* chemotherapy (in the case of nitrosoureas and mitomycin C within 6 weeks), radiotherapy, immunotherapy, or any other study drug within 3 weeks before study drug administration
* antibody based cancer therapy within 4 weeks before administration of the first dose of DO-2
* patients who became progressive on previous treatment with a MET-kinase inhibitor
* patients with brain metastases are excluded unless all of the following criteria are met:

  1. CNS lesions are asymptomatic and previously treated
  2. No ongoing requirement for corticosteroids as therapy for CNS metastases
  3. Imaging demonstrates stability of disease > 28 days from last treatment for CNS metastases
* leptomeningeal involvement (leptomeningeal carcinomatosis)
* history of uncontrolled heart disease including unstable angina, congestive heart failure, myocardial infarction within preceding 12 months, clinically significant rhythm or conduction abnormality, congenital long QT syndrome, obligate use of a cardiac pacemaker, QTc at screening greater than 450 milliseconds in males and greater than 470 milliseconds in females
* uncontrolled arterial hypertension despite appropriate therapy
* positive pregnancy test (urinary beta-hCG) at screening (applicable to women of child-bearing potential who are sexually active)
* mental status alteration or history of major psychiatric illness, which may potentially impair patient's compliance with study procedures
* signs and symptoms of active infection requiring systemic therapy
* other medical condition (e.g. pre-existing kidney dysfunction) that in the opinion of the investigator makes it undesirable for a patient to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects who experience Dose Limiting Toxicities (DLTs) | Baseline up to Week 4
  Only toxicities that occur during Cycle 1 will be considered for the purposes of defining DLT and for dose escalation, but toxicities that occur in all cycles will be recorded and considered in decisions about the Maximum Tolerated Dose. DLTs are defined as toxicities that meet pre-defined severity criteria. Toxicity grading will be performed in accordance with NCI-CTC Version 5.0.
Number of subjects who experience specific treatment-related adverse events (TRAEs) | Baseline up to Week 36
  Number of subjects with specific treatment-related adverse events for each dose group.
  AE refers to any untoward medical occurrence or deterioration of existing medical event after the subject signed the ICF, whether or not considered related to the study treatment. TRAEs are any event that occurs after the subject has received study treatment. AE grading will be performed in accordance with NCI-CTC Version 5.0.
Determination of the Maximum Tolerated Dose (MTD) | Baseline up to Week 4
  The MTD in milligram is defined as the highest dose at which less than one third of the subjects in a dose level cohort experience DLT.

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) and Area under the curve (AUC) of DO-2 | Baseline up to Day 23
  Determine the Cmax and AUC of DO-2 and its main metabolites in plasma sampled at different timepoints during Cycle 1.
Time over treshold (ToT) for DO-2 | Baseline up to Day 23
  Time by which the observed concentration of DO-2 in plasma is above the expected efficacy treshold.
Objective responses seen in Part I and objective response rate (ORR) in Part II | Baseline through study completion, an average of 36 weeks
  ORR is defined as the proportion of subjects with confirmed CR or confirmed PR. Radiologic assessment will be repeated after every second cycle (or more frequently if clinically indicated) and using same methodology as at baseline. Response assessment (radiologic) will be determined in accordance with RECIST (version 1.1) and current disease specific solid tumour response criteria.
Duration of response (DoR) | Baseline through study completion, an average of 36 weeks
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression (based on RECIST Version 1.1) or death due to any cause, whichever occurs first.
Progression-free survival (PFS) | Baseline through study completion, an average of 36 weeks
  PFS is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first (based on RECIST Version 1.1).
Overall survival (OS) | Baseline through study completion, an average of 36 weeks
  OS defined as the time from the first dose to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Verweij, MD, Study Chair — CMO DeuterOncology
Locations (8):
- Belgium (3):
  - Institut Roi Albert II - UC Louvain, Brussels
  - UZA, Edegem
  - Universitair Ziekenhuis Gent, Ghent
- France (3):
  - Centre Georges-François Leclerc - CHU Dijon, Dijon
  - Institut Cœur Poumon - CHU Lille, Lille
  - Centre Léon Bérard, Lyon
- Netherlands (2):
  - Radboud UMC, Nijmegen
  - Erasmus Medical Centre, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: DeuterOncology Internet site — https://www.deuteroncology.com/